CLINICAL TRIAL: NCT01787695
Title: UVA 1 Phototherapy for Vitiligo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H10-02235
Record Dates: First submitted 2013-02-04; First posted 2013-02-11 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Vitiligo
Keywords: Vitiligo; UVA1; Phototherapy
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- No treatment (covered) (No Intervention)
- UVA1 (Active Comparator)
  Interventions: Procedure: UVA1

INTERVENTIONS:
Procedure: UVA1 — Patients with a vitiligo patch larger than 25cm2 will be recruited. The target patch will be divided into two halves. One half will be shielded by foil and served as control while the other half will be exposed to UVA1.
  The dose of UVA1 will be 60 J/cm2, 5 times a week for 4 weeks. Patients that have no or less than 10% pigmentation change after 4 weeks will receive UVA1 130J/cm2, 5 times a week for another 4 weeks. The patients with more than 10% pigmentation change will receive UVA1 60 J/cm2, 5times a week for another 4weeks. This will be followed by assessments at 4, 8, and 12 weeks post treatment.
  Arms: UVA1

SUMMARY:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin. There are many treatment modalities available for vitiligo, however, none of them cure the disease. Ultraviolet A1 (UVA1) phototherapy has been shown to be useful for a variety of skin diseases. However, there are only a few studies published on the efficacy of UVA1 in vitiligo. This is a prospective single-blind randomized clinical trial to assess efficacy and safety of UVA1 in the treatment of vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a chronic acquired disease characterized by well defined white macules and patches affecting the skin and mucous membranes. Mucocutaneous lesions develop secondary to selective destruction of melanocytes. The etiology of vitiligo is largely unknown but more likely to be multifactorial. There are several theories on the pathogenesis of vitiligo including mainly the autoimmune, neurohormonal, and autocytotoxic theories. The autoimmune hypothesis has the strongest evidence with alteration mainly in the cellular immune response.

There are many treatment modalities available for vitiligo, however, none of them cure the disease. These include different topical treatments, phototherapy, surgical therapy, and depigmentation therapy. Narrow-band UVB (NB-UVB) is currently the preferred treatment over topical psoralen and ultraviolet A radiation (PUVA), for patients with vitiligo. However, overall response of vitiligo to NB-UVB has been variable. Ultraviolet A1(UVA1) phototherapy is now useful for a variety of skin diseases, specifically scleroderma. There are only a few studies published on the efficacy of UVA1 in vitiligo.

One of the main side effects of UVA1 is prominent tanning which might be due to melanocyte stimulation. Therefore, the investigators hypothesis is that UVA1 will induce significant skin pigmentation to improve vitiligo. The investigators plan on conducting a prospective single-blind randomized clinical trial to assess efficacy and safety of UVA1 in the treatment of vitiligo.

Study Objectives

1. To evaluate the potential for UVA1 to induce repigmentation within vitiligo patches.
2. To assess the side effect profile of UVA1 when used in the treatment of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Localized or generalized vitiligo that involves a non mucosal or acral site.
* Patients should have a patch of at least 25 cm2 that shows no more than 10% repigmentation as assessed visually

Exclusion Criteria:

* Patients who received treatment for vitiligo within the past 3 weeks.
* Patients known to have a photosensitivity disorder
* History of previous skin cancer.
* History of severe medical illness or immunosuppression.
* Pregnancy or breast-feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in the modified VASI score compared to baseline. | assessments at 2, 4, 6, and 8 weeks during treatment then at 4, 8, and 12 weeks post treatment

SECONDARY OUTCOMES:
Assessment of side effects in each half including erythema, pruritus, and polymorphous light eruption | assessments at 2, 4, 6, and 8 weeks during treatment then at 4, 8, and 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lui, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, British Columbia, Canada